CLINICAL TRIAL: NCT00145067
Title: Three Methods of Delivering Health Care for Secondary Prevention of Osteoporosis
Brief Title: Osteoporosis Disease Management Demonstration Project (0000-040)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0000-040; 040; 2005_051
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

INTERVENTIONS:
Behavioral: Disease Management Assessment

SUMMARY:
The purpose of the study is to evaluate the impact disease management interventions in treatment compliance among post-fracture and osteoporosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Members of of the Kaiser Permanente Health Plan who have fractured a bone.

Exclusion Criteria:

* Individuals who are not members of the Kaiser Permanente Health Plan.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2003-11; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Treatment persistence

SECONDARY OUTCOMES:
Patient satisfaction and knowledge

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Waalen J, Bruning AL, Peters MJ, Blau EM. A telephone-based intervention for increasing the use of osteoporosis medication: a randomized controlled trial. Am J Manag Care. 2009 Aug 1;15(8):e60-70. PMID 19659407